CLINICAL TRIAL: NCT04447521
Title: A 20-months Surveillance of Non-invasive Streptococcus Pneumoniae Infections in Belgium to Evaluate National Vaccination Strategy
Brief Title: Surveillance of Non-invasive Streptococcus Pneumoniae Infections in Belgium
Acronym: STREPTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sciensano (Other Government)
Collaborators: Pfizer (Industry); Merck Sharp & Dohme LLC (Industry); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: STREPTO1.2
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia; Otitis Media; Sinusitis Bacterial
MeSH Terms: conditions — Pneumonia; Otitis Media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Streptococcus pneumoniae samples will be collected and stored during the time frame of this study.
  DNA extraction and whole-genome sequencing will be performed for a subset of these strains.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will conduct a prospective observational study of non-invasive S. pneumoniae infections in Belgium and characterize serotype distributions to evaluate national vaccination programs.

DETAILED DESCRIPTION:
The investigators will conduct a surveillance of non-invasive S. pneumoniae infections in Belgium (September 2020-May 2025). Monthly, 12 peripheral hospitals will send the first 15 unduplicated clinical S. pneumoniae samples (coming from patients diagnosed with pneumonia, otitits media or sinusitis) to the investigators. The investigators will determine the serotype and the antibiotic resistance profile of these clinical isolates. Whole genome sequencing will be performed on a subset of these isolates.

From May 2021, 13 extra participating centers have been added to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients living in Belgium at the time of the study,
* from whom unduplicated S. pneumoniae isolates were collected in routine practices,
* from non-invasive upper (e.g.: pus/fluid from nasal sinus or from otitis media fluid) or lower respiratory tract (e.g. sputum bronchial or endotracheal aspirate, bronchoalveolar fluid (BAL),…) clinical samples,
* from patients diagnosed with pneumonia, sinusitis and otitis.

Exclusion Criteria:

• Patients for whom S. pneumoniae was simultaneously isolated from blood or another usually sterile specimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from non-invasive pneumococcal disease (diagnosed as CAP, sinusitis and otitits media) and living in Belgium at the time of the study.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish insight in serotype dynamics for non-invasive pneumococcal diseases in Belgium prospectively, in association with changing vaccination programs (campaigns). | September 2020-May 2025
  There is a wealth of information available on the serotype distribution of S. pneumoniae causing inavsive pneumococcal disease (IPD). However, much less is known about the serotype distribution of S. pneumoniae causing non-invasive pneumococcal disease (NIPD). The goal of this study is to characterize the serotype distribution of of S. pneumoniae causing NIPD in Belgium, compare is with IPD data and link it with the changing national vaccinations programs.

SECONDARY OUTCOMES:
Surveillance of emerging serotypes, clones and drug resistances. Study of the genetic divergences between invasive and non-invasive pneumococcal diseases isolates. | September 2020-May 2025
  To date, little is known about serotype distribution in NIPD and how this relate with the more widely studied serotype distribution in IPD. This study aims to shed light onto this topic.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter-Jan Ceyssens, PhD, Principal Investigator — Sciensano
Locations (1):
- Sciensano, Brussels, Belgium

DOCUMENTS (1):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04447521/Prot_000.pdf